CLINICAL TRIAL: NCT01588158
Title: Satisfaction With Pain Relief After Carpal Tunnel Release Surgery
Brief Title: Patient Satisfaction With Pain Relief After Ambulatory Hand Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The PI of this study is leaving the institution and enrollment was progressing slowly so we decided to close the study.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Associate Professor of Orthopaedic Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011P001670
Record Dates: First submitted 2012-04-25; First posted 2012-04-30 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; Tylenol; Vicodin; pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain | interventions — Acetaminophen; acetaminophen, hydrocodone drug combination; Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vicodin 5/325 mg (Active Comparator): Half of the patients will be randomized to Vicodin
  Interventions: Drug: Acetaminophen
- Acetaminophen 325 mg (Active Comparator): Half of the patients will be randomized to Acetaminophen
  Interventions: Drug: Vicodin

INTERVENTIONS:
Drug: Acetaminophen — 325 mg
  Other Names: Tylenol
  Arms: Vicodin 5/325 mg
Drug: Vicodin — Vicodin 5/325 mg
  Other Names: Hydrocodon/Acetaminophen
  Arms: Acetaminophen 325 mg

SUMMARY:
Adequate pain relief has been a priority of the Joint Commission and is featured on national inpatient surveys such as the H-CAHPS. When considering methods for improving satisfaction with pain relief in the United States, a great deal of emphasis has been placed on opioid pain medications. Some of this emphasis on opioid pain medication is driven by the pharmaceutical industry and by advocacy groups with ties to the pharmaceutical industry.

There is evidence that the "pain is the fifth vital sign" campaign of the Joint Commission led to an increased incidence of prescription of opioids, but there is less evidence of improved satisfaction with pain relief. There is some evidence of an increase in opioid-related adverse events. As the sales of opioids have tripled from 1999-2008, so has the number of deaths caused by opioid overdose; 14,800 in 2008. The number of visits to the Emergency Department for opioid overdose doubled between 2004 and 2008.

Patients in other countries take far less opioid pain medication and are equally satisfied with pain relief. For instance, Lindenhovius et al. found in a retrospective study that Dutch patients take a weak (Tramadol) or no opioid pain medication after ankle fracture surgery and have comparable or better satisfaction with pain relief than American patients, most of whom take oxycodone. That study was repeated prospectively (unpublished) and confirmed that Dutch patients do not feel their pain is undertreated. A study of morphine use after a femur fracture demonstrated that American patients used far more than Vietnamese patients (30 mg/kg versus 0.9 mg/kg), but were more dissatisfied with their pain relief. These sociological differences are striking and suggest strongly that personal factors may be the most important determinant of satisfaction with pain relief.

It is our impression that most American hand surgeons give patients a prescription for an opioid pain medication after carpal tunnel release, and that is certainly true in our practice. This seems to be based primarily on the outliers, and intended to avoid confrontation with patients that desire opioids; however, most patients take little or no narcotic pain medication, and many who do use the opioids complain of the side effects-nausea and pruritis in particular. It is therefore not clear whether routine opioids is the optimal pain management strategy after carpal tunnel release. In the study of Stahl et al. from Israel, patients were prescribed acetaminophen rather than opioids after carpal tunnel release and only 20 of 50 patients used acetaminophen; 30 patients did not use acetaminophen or other pain medication at all after the operation.

Our aim is to determine if there is a difference in satisfaction with pain relief between patients advised to take opioids compared to patients advised to use over the counter acetaminophen after carpal tunnel release under local anesthesia. A secondary aim is to determine if personal factors account for more of the variability in satisfaction with pain relief than opioid strategy.

DETAILED DESCRIPTION:
Aim:

The specific aim of this study is to compare the effectiveness of Tylenol and Vicodin after carpal tunnel release.

Primary Study Question:

There is no difference in satisfaction with pain relief at the time of suture removal between those advised to use acetaminophen instead of opioids and those give standard advice and a standard prescription for opioids.

Secondary Study Questions/Null Hypotheses:

1. Psychological and demographic factors do not account for variation in satisfaction with pain relief.
2. Arm-specific disability does not correlate with use of opioid pain medication.
3. Overall pain during recovery does not correlate with use of opioid pain medication.

Adequate pain relief has been a priority of the Joint Commission and is featured on national inpatient surveys such as the H-CAHPS. When considering methods for improving satisfaction with pain relief in the United States, a great deal of emphasis has been placed on opioid pain medications. Some of this emphasis on opioid pain medication is driven by the pharmaceutical industry and by advocacy groups with ties to the pharmaceutical industry. For instance 88% of the income of the American Pain Foundation is from industry. It is a consistent finding that although opioid pain improves pain in comparison with placebo, there is no difference in disability or pain relief compared to NSAIDs.

There is evidence that the "pain is the fifth vital sign" campaign of the Joint Commission led to an increased incidence of prescription of opioids, but there is less evidence of improved satisfaction with pain relief. There is some evidence of an increase in opioid-related adverse events. As the sales of opioids have tripled from 1999-2008, so has the number of deaths caused by opioid overdose; 14,800 in 2008. The number of visits to the Emergency Department for opioid overdose doubled between 2004 and 2008.

Patients in other countries take far less opioid pain medication and are equally satisfied with pain relief. For instance, Lindenhovius et al. found in a retrospective study that Dutch patients take a weak (Tramadol) or no opioid pain medication after ankle fracture surgery and have comparable or better satisfaction with pain relief than American patients, most of whom take oxycodone. That study was repeated prospectively (unpublished) and confirmed that Dutch patients do not feel their pain is undertreated. A study of morphine use after a femur fracture demonstrated that American patients used far more than Vietnamese patients (30 mg/kg versus 0.9 mg/kg), but were more dissatisfied with their pain relief. These sociological differences are striking and suggest strongly that personal factors may be the most important determinant of satisfaction with pain relief.

It is our impression that most American hand surgeons give patients a prescription for an opioid pain medication after carpal tunnel release, and that is certainly true in our practice. This seems to be based primarily on the outliers, and intended to avoid confrontation with patients that desire opioids; however, most patients take little or no narcotic pain medication, and many who do use the opioids complain of the side effects-nausea and pruritis in particular. It is therefore not clear whether routine opioids is the optimal pain management strategy after carpal tunnel release. In the study of Stahl et al. from Israel, patients were prescribed acetaminophen rather than opioids after carpal tunnel release and only 20 of 50 patients used acetaminophen; 30 patients did not use acetaminophen or other pain medication at all after the operation.

Our aim is to determine if there is a difference in satisfaction with pain relief between patients advised to take opioids compared to patients advised to use over the counter acetaminophen after carpal tunnel release under local anesthesia. A secondary aim is to determine if personal factors account for more of the variability in satisfaction with pain relief than opioid strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* All subjects will be competent adults able to consent on their own behalf for surgery and care.
* Inclusion prior to surgery
* Carpal tunnel release

Exclusion Criteria:

* Pregnant women. Patients will be queried with the routine preoperative medical history and an inclusion/exclusion checklist.
* Patients unable to give informed consent
* Non English-speaking subjects
* Patients with hypersensitivity to acetaminophen or hydrocodone
* Patients with chronic alcohol abuse
* Patients with severe impairment of renal or hepatic function. This will be assessed in the routine preoperative medical history and review of the medical record. We will also ask the patients specific for this history in the screening for the study inclusion/exclusion criteria.
* Patients with hypothyroidism
* Patients with Addison's disease
* Patients with prostatic hypertrophy or urethral stricture
* Patients using any of the following medications:

MAO or tricyclic antidepressants Antihistaminics Antipsychotic or anti-anxiety medications Phenothiazines Zidovudin Phenobarbital

* Patients who are taking opioid pain medication for another reason prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Ring, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (7.5) | 50 (13.1) | 57.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Pain Relief
Description: an 11-point ordinal scale to ask for the satisfaction of the patients with pain relief. The scale range is from 0-10, where 0 is complete dissatisfaction with pain relief and 10 is complete satisfaction.
Time Frame: at the follow-up, 2 weeks after the operation with suture removal
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Number analyzed (Participants) | 4 | 3
units on a scale | 6.75 (2.75) | 6.67 (5.77)

2. Secondary Outcome: QuickDASH
Description: The short form of the Disabilities of Arm Shoulder and Hand to assess upper extremity disability. The scale range is from 0-100, where 0 is no difficulty performing tasks and 100 is the most difficulty or unable to complete any tasks.
Time Frame: At enrollment prior to surgery
Population: Due to early termination of the study, the participants were not analyzed so we do not have data to enter in the outcome measure data table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Number analyzed (Participants) | 4 | 3
units on a scale | 41.5 (19.51) | 33.3 (9.46)

3. Secondary Outcome: PSEQ
Description: The pain self efficacy questionnaire measures a patient's belief about his/her ability to complete a task despite his/her pain. The scale range is from 0-60, where 60 represents higher self-efficacy beliefs.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Number analyzed (Participants) | 4 | 3
units on a scale | 41.75 (19.10) | 46 (8.7)

4. Secondary Outcome: PHQ-9
Description: Patient Health Questionnaire-9 to assess symptoms of depression. The scale range is from 0-27, where 0 is no symptoms of depression and 27 is severe depression.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Number analyzed (Participants) | 4 | 3
units on a scale | 6.5 (5.2) | 4.7 (4.2)

5. Secondary Outcome: Pain Patients Expect After Surgery
Description: an 11-point ordinal scale to assess the amount of pain the patients expect after surgery. The scale range is from 0-10, where 0 is no pain expected and 10 is the worst pain expected
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Number analyzed (Participants) | 4 | 3
units on a scale | 3.5 (1.73) | 4 (2.65)

6. Secondary Outcome: Expectation of Pain Relief
Description: An 11-point ordinal scale to assess the expectation of how well the pain medication will work after surgery. The scale range is from 0-10, where 0 is not effective at all and 10 is completely effective.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Number analyzed (Participants) | 4 | 3
units on a scale | 8.25 (0.5) | 8.33 (1.53)

7. Secondary Outcome: Pain Scale
Description: 11-point ordinal pain scale to assess the amount of pain. The scale range is from 0-10, where 0 is no pain at all and 10 is the worst pain ever had.
Time Frame: At enrollment prior to surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Number analyzed (Participants) | 4 | 3
units on a scale | 4.75 (2.5) | 6 (2)

8. Secondary Outcome: QuickDASH
Description: as for outcome 2
Time Frame: At the follow-up 2 weeks after the surgery with suture removal
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Number analyzed (Participants) | 4 | 3
units on a scale | 46.0 (19.9) | 36.4 (35)

9. Secondary Outcome: Pain Scale
Description: as for outcome 7
Time Frame: At the follow-up 2 weeks after the surgery with suture removal
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Number analyzed (Participants) | 4 | 3
units on a scale | 4.5 (4.12) | 1.3 (2.3)

ADVERSE EVENTS:
Time Frame: 3 years, 9 months
Arm/Group | Vicodin 5/325 mg | Acetaminophen 325 mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No